CLINICAL TRIAL: NCT03912389
Title: International Multicenter Randomized Double-Blind Placebo-Controlled Clinical Trial Evaluating Efficacy and Safety Of BCD-100 in Combination With Pemetrexed+Cisplatin/Carboplatin Compared to Placebo in Combination With Pemetrexed+Cisplatin/Carboplatin as First-Line Treatment of Subjects With Advanced Non-squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Efficacy and Safety of BCD-100 (Anti-PD-1) in Combination With Platinum-Based Chemotherapy as First Line Treatment in Patients With Advanced Non-Squamous NSCLC
Acronym: DOMAJOR
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-100-3
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Non-Squamous Non-Small Cell Neoplasm of Lung
MeSH Terms: interventions — Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-100 (Experimental): BCD-100 3 mg/kg Q3W
  Interventions: Biological: BCD-100; Drug: Pemetrexed; Drug: Cisplatin (or carboplatin)
- Placebo (Placebo Comparator)
  Interventions: Drug: Pemetrexed; Drug: Cisplatin (or carboplatin); Other: Placebo

INTERVENTIONS:
Biological: BCD-100 — Anti-PD-1 monoclonal antibody, IV infusion
  Arms: BCD-100
Drug: Pemetrexed — IV infusion
Drug: Cisplatin (or carboplatin) — IV infusion
Other: Placebo — IV infusion
  Arms: Placebo

SUMMARY:
This is a randomized, multicenter, double-blind placebo-controlled phase 3 study of efficacy and safety of BCD-100 in combination with pemetrexed+cisplatin/carboplatin compared to placebo in combination with pemetrexed+cisplatin/carboplatin in subjects with previously untreated metastatic non-squamous NSCLC. The main hypothesis of the study is that BCD-100 in combination with chemotherapy prolongs OS compared to placebo with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has voluntarily agreed to participate by giving written informed consent for the trial;
2. Patients ≥ 18 years of age on day of signing informed consent;
3. Previously untreated patients with histologically-confirmed stage IV (M1a/M1b/M1c- AJCC 8th edition) non-squamous NSCLC;
4. Has not received prior systemic treatment for metastatic NSCLC;
5. The time from the completion of previous adjuvant/neoadjuvant treatment to metastatic disease development is no less than 12 months;
6. Has a life expectancy of at least 12 weeks;
7. Has Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1;
8. Has adequate organ function as defined by hematological laboratory values (absolute neutrophil count ≥1.500/mcL, platelets ≥100.000/mcL, hemoglobin ≥9 g/dL ), renal laboratory values (serum creatinine or calculated creatinine clearance <1.5xULN or ≥60 mL/min for subjects with creatinine levels>1.5x institutional ULN), and hepatic laboratory values (serum total bilirubin <1.5xULN, AST and ALT ≤2.5xULN, alkaline phosphatase <2.5xULN);
9. Agreement to newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for determination of PD-L1 status prior to randomization (if obtaining of new sample is contraindicated or puts subject at unacceptable risks, then archival tumor tissue sample must be available)
10. Measurable disease according to CT scan (RECIST 1.1 criteria) , confirmed by the local assessment;
11. For subjects of childbearing potential: agreement to remain abstinent (refrain from heterosexual inter-course) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 6 months after administration of the last dose of study drug; and 6 months after the last dose of platinum-based chemotherapy, whichever is later. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes, and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include but are not limited to bilateral tubal ligation and/or occlusion, male sterilization, and intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

1. Has predominantly squamous cell histology NSCLC; Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the subject is ineligible.
2. Presence of EGFR mutation or ALK translocation;
3. Has received prior systemic cytotoxic chemotherapy/chemoradiotherapy for metastatic disease;
4. Has received antineoplastic therapy with targeted or immunotherapeutic drugs (including but not limited to EGFR inhibitors [e.g., erlotinib, gefitinib, cetuximab], ALK inhibitors, PD-1/PD-L1/PD-L2/CTLA4, VEGF/VEGFR inhibitors) or it is expected to require any other form of antineoplastic therapy while on study;
5. Completed radiation therapy within 14 days before the first dose of the study drug;
6. Received a live-virus vaccination within 30 days prior to the first study drug administration;
7. Current treatment in another investigational device or drug study, or less than 28 days since ending treatment on another investigational device or drug study;
8. Had major surgery less than 28 days prior to the first dose of the study drug;
9. Evidence of severe or concomitant diseases/life-threatening complications of the main condition (including but not limited to massive pleural, pericardial, or peritoneal effusion that requires medical intervention , pulmonary lymphangitis, hemorrhage, organ perforation) at the signing of the informed consent;
10. Concomitant diseases or conditions which pose a risk of AE development during study treatment:

    1. uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg; define diagnosis of hypertension
    2. stable angina functional class III-IV;
    3. unstable angina or myocardial infarction less than 6 months prior to randomization;
    4. NYHA Grade III-IV congestive heart failure;
    5. serious cardiac arrhythmia requiring medication (subjects with asymptomatic atrial fibrillation can be enrolled if controlled ventricular rate);
    6. atopic asthma, Stage III-IV COPD, angioedema;
    7. severe respiratory failure;
    8. any other diseases which pose unacceptable risk of AE development during study treatment in Investigator's opinion;
11. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis ;
12. Active or known or suspected autoimmune disease (subjects with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, or skin disorders (vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll).
13. Has clinically active diverticulitis, intra-abdominal abscess, GI obstruction, abdominal carcinomatosis;
14. Has interstitial lung disease or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management. Lymphangitic spread of the NSCLC is not exclusionary;
15. Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications in past 2 years;
16. Is unable or unwilling to take folic acid or vitamin B12 supplementation;
17. Known history of prior malignancy except if participant has undergone potentially curative therapy with no evidence of that disease recurrence for 2 years since initiation of that therapy, except for successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers;
18. Pre-existing clinically significant (≥ grade 2) peripheral neuropathy or hearing impairment;
19. Any conditions or circumstances that limit subject's ability to comply with protocol requirements;
20. Active hepatitis B, hepatitis С or HIV in anamnesis;
21. Acute infection or reactivation of chronic infection or systemic antibiotics use less than 14 days prior to first dose of the study drug; Severe infections within 28 days prior to the first study drug administration.
22. Significant adverse reactions of previous therapy excluding chronic and/or irreversible events which cannot affect study drug safety evaluation (e.g. alopecia);
23. Known hypersensitivity or allergy to drugs containing Chinese hamster (CHO) ovary cells or history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, to pemetrexed, carboplatin, cisplatin, BCD-100 or any of their excipients;
24. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3 years
  The time from the date of randomization until death

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 1 year
  The time from the date of randomization until progression of disease according to RECIST 1.1 and iRECIST or death
Overall Response Rate (ORR) | 1 year
  The percentage of the participants who have a Complete Response or a Partial Response as assessed by a blind independent central reviewer per RECIST 1.1 and iRECIST
Disease Control Rate (DCR) | 1 year
  The percentage of the participants who have a Complete Response, a Partial Response or a Stable Disease as assessed by a blind independent central reviewer per RECIST 1.1 and iRECIST
Time to Response (TTR) | 1 year
  TTR will be calculated from the randomization date
Duration of Response (DOR) | 1 year
  DOR will be calculated from the moment of registration of response till event (disease progression or death)

CONTACTS AND LOCATIONS:
Overall Officials: Yulia N Linkova, MD, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (37):
- Czechia (4):
  - Regional Hospital Liberec, Liberec
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - Multiscan Pardubice - Radiology Center, Pardubice
- Georgia (5):
  - High technology Hospital Medcenter, Batumi
  - Acad. F.Todua Medical center "Research institute of Clinical Medicine", Tbilisi
  - High Technology Medical Centre, University Clinic, Tbilisi
  - Institute for Personalized Medicine Ltd., Tbilisi
  - LEPL First University Clinic of Tbilisi State Medical University, Tbilisi
- Hungary (3):
  - National Korányi Institute of Pulmonology IV. Pulmonology, Budapest
  - Semmelweis University Pulmonology Clinic, Budapest
  - Mátra Health Institution Pulmonology, Mátraháza
- Romania (9):
  - S.C Medisprof S.R.L, Cluj-Napoca
  - S.C Radiotherapy Center Cluj S.R.L, Cluj-Napoca
  - "Sfantul Nectarie" Oncology Center SRL, Craiova
  - S.C Oncolab S.R.L, Craiova
  - S.C Pelican Impex S.R.L, Oradea
  - Emergency Clinical Municipal Hospital Timisoara - Medical Oncology Clinic, Timișoara
  - S.C Oncocenter Clinical Oncology S.R.L, Timișoara
  - S.C Oncomed S.R.L, Timișoara
  - S.C Salvosan Ciobanca S.R., Zalău
- Russia (9):
  - Arkhangelsk Clinical Oncology Dispensary, Arkhangelsk
  - City Hospital No. 5, Barnaul
  - Krasnoyarsk Regional Clinical Oncological Dispensary named after A.I. Kryzhanovsky, Krasnoyarsk
  - Moscow City Oncology Hospital No. 62, Moscow
  - Clinical Oncology Dispensary, Omsk
  - LLC "New Clinic", Pyatigorsk
  - AV Medical Group, Saint Petersburg
  - LLC BioEk, Saint Petersburg
  - Regional Clinical Oncology Hospital, Yaroslavl
- Slovakia (7):
  - St. Jacob's Hospital, Bardejov
  - Hospital Komarno a.s., Komárno
  - Eastern Slovak Oncology Institute, Košice
  - Faculty Hospital with Policlinic of Stefan Kukura, Michalovce
  - Faculty Hospital with Policlinic, Nové Zámky
  - Outpatient Oncology Clinic, Partizánske
  - Faculty Hospital of J.A. Reiman, Prešov

REFERENCES:
- [Derived] Laktionov K, Smolin A, Stroyakovskiy D, Moiseenko V, Dvorkin M, Andabekov T, Cheng Y, Liu B, Kozlov V, Odintsova S, Dvoretsky S, Mochalova A, Urda M, Yi T, Li X, Laszlo U, Muller V, Bogos K, Fadeeva N, Musaev G, Liu Q, Kirtbaya D, Shi J, Gladkov O, Narimanov M, Semiglazova T, Khasanova A, Chovanec J, Andrasina I, Szabova A, Rosinska O, Sudekova D, Zsolt PS, Ran F, Sun M, Jiang O, Chen R, Zhao E, Liu C, Tan W, Pirmagomedov A, Poddubskaya E, Kislov N, Shumskaya I, Sorokina I, Zinkina-Orikhan A, Linkova Y, Fogt S, Liaptseva D, Siliutina A, Basova O, Kryukov F. Prolgolimab with chemotherapy as first-line treatment for advanced non-squamous non-small-cell lung cancer. Eur J Cancer. 2025 Feb 25;217:115255. doi: 10.1016/j.ejca.2025.115255. Epub 2025 Jan 21. PMID 39879779